CLINICAL TRIAL: NCT03243513
Title: Abortion Follow-up Study
Brief Title: Abo Follow-up Study
Status: Terminated | Type: Observational
Why Stopped: PI has confirmed that this is not a clinical trial and was entered in error in the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Lisa Hofler, Assistant Professor, University of New Mexico
Other Study IDs: 17-276
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Termination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective Chart Review — There is no intervention in this research. This research project is a retrospective chart review.

SUMMARY:
The aim of the project is to identify an efficient and effective policy or procedure for identifying complications from surgical abortions through follow-up phone calls.

DETAILED DESCRIPTION:
The aim of the project is to identify an efficient and effective policy or procedure for identifying complications from surgical abortions through follow-up phone calls. Key questions include, what is our complication-detection rate from these phone calls? How many patients are contacted? How many attempts are made and how much effort is expended by staff in routine follow-up practices? Additionally, the research would attempt to answer the question, is there any way to predict problems or complications? This study will help to determine if excessive resources and time are being expended on follow-up phone method to detect complications.

This study will consist of a retrospective chart review identifying the outcome of follow-up phone calls after an induced abortion.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive-aged women
* women who have had an induced abortion, and are contacted by a clinical nurse for a follow-up phone call.

Exclusion Criteria:

-

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: De-identified charts of women who have had an induced abortion and are contacted by a nurse for a follow-up phone call.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Follow-up Phone Calls | 2 years
  Key questions include, what is our complication-detection rate from these phone calls? How many patients are contacted? How many attempts are made and how much effort is expended by staff in routine follow-up practices?

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hofler, MD, MBA, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing IPD at this time